CLINICAL TRIAL: NCT00004017
Title: Phase II Open-Label, Non-Randomized, Multicenter Study of Interstitial 131I-chTNT-1/B for the Treatment of Newly Diagnosed or Recurrent Malignant Glioma
Brief Title: Radiolabeled Monoclonal Antibody in Treating Patients With Glioblastoma Multiforme or Anaplastic Astrocytoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peregrine Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067235; PEREGRINE-TNT9802; MUSC-7993; PEREGRINE-BB-IND-7344; TCLONE-BB-IND-7344; TCLONE-TNT9802; NCI-G99-1560
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2003-03

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Gliosarcoma | interventions — 131I-chimeric TNT-1-B monoclonal antibody

INTERVENTIONS:
Procedure: conventional surgery
Radiation: iodine I 131 monoclonal antibody TNT-1/B

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies can locate tumor cells and deliver tumor-killing substances to them without harming normal cells. This may be an effective treatment for some types of brain tumors.

PURPOSE: Phase II trial to study the effectiveness of radiolabeled monoclonal antibody in treating patients who have glioblastoma multiforme or anaplastic astrocytoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the median time to disease progression in patients with newly diagnosed unresectable glioblastoma multiforme (GBM), recurrent GBM, or recurrent anaplastic astrocytoma treated with interstitial iodine I 131 monoclonal antibody TNT-1/B.
* Determine the median survival time of these patients treated with this regimen.
* Determine the safety of this regimen in terms of neurotoxicity, renal, hepatic, hematologic, and biochemical profiles in these patients.
* Confirm the maximum tolerated dose of this regimen in these patients.
* Optimize the drug delivery of this regimen in these patients.
* Assess the response of these patients in terms of MRI measured gadolinium enhanced tumor volume and gadolinium enhanced tumor area at 8 and 12 weeks following the last dose of study drug.

OUTLINE: This is a multicenter study.

Patients undergo stereotactic implantation of 2 interstitial catheters into the tumor bed. One day later, patients receive iodine I 131 monoclonal antibody TNT-1/B interstitially over approximately 24 hours. At selected centers, up to 3 additional groups of 3 patients each will receive study drug up to 48 hours. Catheters are removed 1 day after completion of the infusion. A gadolinium enhanced MRI is performed during week 8. Patients with partial response, minimal response, or stable disease repeat the above treatments during week 9. Patients with complete response, progressive disease, or unacceptable toxicity receive no additional treatment.

Patients are followed every month until disease progression. All patients regardless of disease progression or retreatment are followed at 36 weeks.

PROJECTED ACCRUAL: A total of 60 patients (20 patients with newly diagnosed unresectable glioblastoma multiforme [GBM]; 20 patients with recurrent GBM; and 20 patients with recurrent anaplastic astrocytoma) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed unresectable glioblastoma multiforme (GBM), recurrent GBM, or recurrent anaplastic astrocytoma (AA)
* MRI scan documenting gadolinium enhanced tumor volume of at least 5 cm3, but no greater than 60 cm^3

  * Recurrent GBM and AA must be documented by MRI after the most recent treatment and before any planned surgical debulking
* At least 5 days since prior surgical debulking
* No planned resection of newly diagnosed GBM before or during study
* No bilateral noncontiguous gadolinium enhancing tumors
* No satellite lesions greater than 1.5 cm from anticipated location of interstitial catheter tip
* No more than 2 satellite lesions

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count at least 100,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* WBC at least 3,000/mm^3

Hepatic:

* Hepatitis B surface antigen negative
* Bilirubin no greater than 2.5 times upper limit of normal (ULN)
* SGOT and SGPT no greater than 3 times ULN
* Alkaline phosphatase no greater than 3 times ULN
* Lactic dehydrogenase no greater than 3 times ULN
* Prothrombin time no greater than 1.5 times ULN

Renal:

* Creatinine clearance at least 50 mL/min

Cardiovascular:

* No significant unstable cardiovascular disease
* No New York Heart Association class III/IV heart disease
* No evidence of myocardial infarction within the past 3 months

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* Human antichimeric antibody (HACA) titer no greater than 48 ng/mL
* No anatomical or physiological considerations that would preclude study participation
* No active autoimmune disease, active infection, or traumatic injury requiring treatment
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior intravenous chemotherapy or Gliadel wafers

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 8 weeks since prior external beam or gamma knife radiotherapy

Surgery:

* See Disease Characteristics

Other:

* At least 30 days since prior investigational treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2000-02

CONTACTS AND LOCATIONS:
Overall Officials: Terrence G. Chew, MD, Study Chair — Peregrine Pharmaceuticals
Locations (4):
- United States (4):
  - Carolina Neurosurgery and Spine Associates, Charlotte, North Carolina
  - Temple University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Huntsman Cancer Institute, Salt Lake City, Utah